CLINICAL TRIAL: NCT01348802
Title: A Randomized Trial Comparing "Push" Versus "Pull" Technology for Mobilizing Pain Evidence Into Practice Across Different Health Professions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Joy MacDermid, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: CIHR-228972
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Knowledge Translation; Push-out Evidence; Technology-Based Knowledge Translation; Pain; Interdisciplinary; Physician; Rehabilitation; Nursing; Knowledge Uptake
MeSH Terms: conditions — Pain | interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Push + Pull (Experimental): Push + Pull is evidence on pain that is extracted from medical, nursing, psychology and rehabilitation journals, appraised for quality and relevance, and delivered to clinicians by e-mail alerts or available for searches of the accumulated database.
  Interventions: Behavioral: Push + Pull
- Pull (Placebo Comparator): Pull will be an intervention with a similar front-face but requires clinicians to go to the site and extract evidence from an electronic database.
  Interventions: Behavioral: Pull

INTERVENTIONS:
Behavioral: Push + Pull — Push + Pull is evidence on pain that is extracted from medical, nursing, psychology and rehabilitation journals, appraised for quality and relevance, and delivered to clinicians by e-mail alerts or available for searches of the accumulated database.
  Arms: Push + Pull
Behavioral: Pull — Pull will be an intervention with a similar front-face but requires clinicians to go to the site and extract evidence from an electronic database.
  Arms: Pull

SUMMARY:
Pain is a problem for many Canadians. Unfortunately, many doctors, nurses, therapists, and psychologists have trouble keeping up to date and applying the latest research that might help patients suffering with pain. This study will determine whether sending alerts about new pain research directly to these health professionals, and providing them with access to accumulated alerts, will help. The study will compare knowledge and decisions made by health professionals about managing pain problems. The investigators will compare physicians, nurses, rehab therapists and psychologists at the beginning of the study and after having access to different ways to find out about new pain research. One group will receive alerts about new pain studies that have been found to be high quality and relevant to patient care, and will be able to search the alerts database. The other group will be able to find the same studies,but must go to the database of research studies to locate them. The investigators will include 670 doctors, nurses, rehab therapists, and psychologists in this study. A process like tossing a coin will determine which way they are able to get pain research information. The investigators will monitor how much information they access and how they apply it to managing pain problems. The investigators expect that reminding health care providers about new research findings directly will help them, since difficulty finding studies and lack of time prevent them from using the latest research. The investigators expect that reminders about the latest research will help them make better decisions about caring for patients' pain.

DETAILED DESCRIPTION:
The Problem: Pain affects all Canadians during acute injury or disease. Chronic noncancer pain affects 29% of Canadians, half of whom are unable to participate in their usual work/social roles. Pain is the primary reason that patients consult health practitioners. Research has shown the benefits, harms, and costs of numerous interventions for pain, but uptake of this knowledge is far from satisfactory. Optimizing pain care requires ready access and use of best evidence within and across different disciplines and settings.

The Research Question: The purpose of this randomized trial is to determine whether a technology-based "push" of new, high-quality pain research to physicians, nurses, rehabilitation and psychology professionals results in better knowledge and clinical decision-making around pain, when offered in addition to traditional "pull" evidence technology. A secondary objective is to identify disciplinary variations in response to evidence and differences in the patterns of accessing research evidence.

The Study Sample: 670 Physicians, nurses, occupational/physical therapists and psychologists ((80/group X 2 comparison groups X 4 disciplines) + 30 for dropouts)will be recruited through professional associations, websites/conferences and social media. This provides > 90% power to detect main effects; 80% power for subgroup effects.

Outcome Measures: The primary outcomes are uptake and application of evidence. Uptake will be determined by embedded tracking of what research is accessed during use of the intervention. A random subset of 30 participants/discipline will undergo chart-stimulated recall (CSR) to assess the nature and depth of evidence utilization in actual case management (0, 9 months). A different random subset of 30 participants/discipline will be tested for their skills in accessing evidence using a standardized simulation test (final 3 months). Secondary outcomes include usage and self-reported evidence-based practice attitudes and behaviours (0, 3, 9, 15, 18 months).

Intervention/Methods: Participants who agree to this study of a free literature service will be randomly allocated to Push + Pull versus Pull evidence support. Push + Pull is evidence on pain that is extracted from medical, nursing and rehabilitation journals and appraised for quality and relevance and sent out to clinicians (derived from the successful MacPLUS/Evidence Updates), delivered by e-mail alerts or available for searches of the accumulated database). Pull will be an intervention with a similar front-face but requires clinicians to go to the site and extract evidence from an electronic database. The trial will begin with a 3-month (repeated) baseline, during which average participant use of the standard PULL resource will be monitored. Participants will then be randomly allocated to receive PUSH + PULL or continue to use the PULL resource. After six months, participants will cross over to the alternate intervention for an additional six months. To complete the trial, both groups will finish with three months of PUSH + PULL access.

Analyses: The investigators will use an analysis of covariance (ANCOVA), where discipline and setting are covariates to assess differential responses across main effects of Push + Pull vs. Pull. Content analysis of the CSR interview will be use to describe the application of evidence within actual cases.

Impact/Timeliness: The trial will inform our understanding on information preferences and behaviours across disciplines/practice settings. If this intervention is effective, sustained support will come through professional/health system initiatives emerging to optimize pain management in Canada.

ELIGIBILITY:
Inclusion Criteria:

* licensed physicians, nurses, occupational therapists (OT), physical therapists (PT), or psychologists who see patients at least 1 day/week;
* fluent in English;
* have access to a computer at home or at work which has unrestricted access to the World Wide Web,
* have an active email account

Exclusion Criteria:

* currently participating in other knowledge translation interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Application of evidence (chart-stimulated recall) | 0, 9 months
  A random subset of 30 participants/discipline will undergo chart-stimulated recall to assess the nature and depth of evidence utilization in actual case management.
Skill at accessing research evidence | 15 months
  A different random subset of 30 participants/discipline will be tested for their skills in accessing evidence using a standardized simulation test.

SECONDARY OUTCOMES:
Usage of PainPLUS | Every month
  Embedded tracking of number/frequency of article access and type of evidence. Level of satisfaction with PainPLUS
Attitudes about Evidence-Based Practice Questionnaire | 0, 3, 9, 15, and 18 months
  Knowledge/Attitude/Behaviour Questionnaire
Familiarity/Access to Technology | 0 months

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDermid, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] MacDermid JC, Law M, Buckley N, Haynes RB. "Push" versus "Pull" for mobilizing pain evidence into practice across different health professions: a protocol for a randomized trial. Implement Sci. 2012 Nov 24;7:115. doi: 10.1186/1748-5908-7-115. PMID 23176444
- [Derived] Arumugam V, MacDermid JC, Walton D, Grewal R. The yield and usefulness of PAIN+ and PubMed databases for accessing research evidence on pain management: a randomized crossover trial. Arch Physiother. 2021 Apr 1;11(1):9. doi: 10.1186/s40945-021-00100-7. PMID 33789739
- See also: Protocol published in Implementation Science — http://www.implementationscience.com/content/7/1/115